CLINICAL TRIAL: NCT02772926
Title: Benfotiamine Effect on Advanced Glycation End Products(AGEs) and Soluble Receptors for AGEs(sRAGE) in Type 2 Diabetes Mellitus.
Brief Title: Benfotiamine Effect on Advanced Glycation End Products(AGEs) and Soluble Receptor for AGEs(sRAGE) in Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Claudia Luévano-Contreras, Professor, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIBIUG-P-27-2015
Record Dates: First submitted 2016-04-26; First posted 2016-05-16 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Benfotiamine; Advanced glycation end products; Soluble receptor for AGEs; Endogenous secretory receptor for AGEs
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — benphothiamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 450 g per pill, 2 pills per day to get 900 mg per day
  Interventions: Dietary Supplement: Placebo
- Benfotiamine (Active Comparator): Benfotiamine (S-Benzoylthiamine O-monophosphate) 450 mg per pill, 2 pills per day to get 900 mg per day
  Interventions: Dietary Supplement: Benfotiamine

INTERVENTIONS:
Dietary Supplement: Benfotiamine — Benfotiamine (S-Benzoylthiamine O-monophosphate) 900 mg per day
  Arms: Benfotiamine
Dietary Supplement: Placebo — Placebo 900 mg per day
  Arms: Placebo

SUMMARY:
Several mechanisms have been implicated in the pathophysiology of the complications of diabetes mellitus (DM), one of them is the formation and accumulation of a heterogeneous group of compounds called advanced glycation end products (AGEs). The interaction of these compounds with their receptor, the receptor for advanced glycation end products (RAGE) triggers several signalling pathways which will lead to increase in inflammatory molecules and enhanced reactive oxygen species. In addition, to the membrane receptor RAGE, there are two soluble forms, the soluble RAGE (sRAGE) and the endogenous secretory RAGE (esRAGE), these soluble receptors are capable to bind AGEs and block the AGE-RAGE axis. It has been observed that in diabetes the needs of thiamine are increased, and it could be an inhibition of the pentose phosphate pathway (thiamine is an essential cofactor in this pathway) and activation of other metabolic pathways among them AGEs formation. It has been proposed that supplementation of benfotiamine could decreased the risk of micro and macrovascular complications, and this could be in part because a decreased in the formation of AGEs. For this reason, the objective of this study was to evaluate the effect of benfotiamine on AGEs and its soluble receptors (sRAGE) in patients with type 2 diabetes.

The specific objectives in the current study are:

1. To evaluate and compare clinical and anthropometric characteristics in type 2 DM patients with and without benfotiamine treatment.
2. To evaluate and compare in type 2 DM patients with and without benfotiamine treatment the following biochemical parameters: total AGEs, Carboxymethyl-lysine (CML), sRAGE, glucose, hemoglobin A1c, lipids (total cholesterol, C-HDL, C-LDL, and triglycerides).
3. To evaluate and compare dietary data such as dietary AGEs and macro and macronutrients in type 2 DM patients with and without benfotiamine treatment.

Type of study: This is a randomized, controlled, double-blind clinical trial

Methods 34 patients will be recruited, 17 per group. After signing the inform consent subjects will be assessed for inclusion criteria. Subjects meeting the inclusion criteria and those whom accept to participate will be randomized to receive either a placebo or benfotiamine treatment for 12 weeks.

At the end of the 12 weeks all the basal assessments will be repeated.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) and its related complications are an increasing health burden all over the world. Insulin deficiency or the insulin resistance in patients with diabetes triggers hyperglycemia which is the main responsible for the micro and macrovascular complications. Several mechanisms have been implicated in the pathophysiology of these complications, one of them is the formation and accumulation of a heterogeneous group of compounds called advanced glycation end products (AGEs). The interaction of these compounds with their receptor, the receptor for advanced glycation end products (RAGE) triggers several signalling pathways which will lead to increase in inflammatory molecules and enhanced reactive oxygen species. In addition, to the membrane receptor RAGE, there are two soluble forms, the soluble RAGE (sRAGE) and the endogenous secretory RAGE (esRAGE), these soluble receptors are capable to bind AGEs and block the AGE-RAGE axis. It has been observed that in diabetes the needs of thiamine are increased, and it could be an inhibition of the pentose phosphate pathway (thiamine is an essential cofactor in this pathway) and activation of other metabolic pathways among them AGEs formation.

It has been proposed that supplementation of benfotiamine could decreased the risk of micro and macrovascular complications, here we proposed that this could be because a decreased in the formation of AGEs. For this reason, the objective of this study was to evaluate the effect of benfotiamine on AGEs and its soluble receptors (sRAGE) in patients with type 2 diabetes.

The specific objectives in the current study are:

1. To evaluate and compare clinical and anthropometric characteristics in type 2 DM patients with and without benfotiamine treatment.
2. To evaluate and compare in type 2 DM patients with and without benfotiamine treatment the following biochemical parameters: Carboxymethyl-lysine (CML)(a marker for AGEs levels), sRAGE, glucose, hemoglobin A1c, lipids (total cholesterol, C-HDL, C-LDL, and triglycerides).
3. To evaluate and compare dietary data such as dietary AGEs and macro and macronutrients in type 2 DM patients with and without benfotiamine treatment.

Type of study: This is a randomized, controlled, double-blind clinical trial

Methods 34 patients will be recruited, 17 per group, level of significance is 0.05 and power 80%. Size was calculated by difference in group means divided by standard deviation.

After signing the inform consent subjects will be assessed for inclusion criteria. Subjects meeting the inclusion criteria and those whom accept to participate will be randomly assigned to receive either a placebo or benfotiamine treatment for 12 weeks. The randomization will be done with a statistical Software (SPSS, V. 21, Chicago).

After group assignment, subjects will be instructed to assist to the Research Center three times for initial assessments.

During the first visit the subject will answer a questionnaire with personal data, medical history and current medications. Patients will be asked to have 10-12 hours of fasting for the blood sample and for the body composition assessment, weight, height and waist circumference will be measured too. Also the blood pressure will be measured during this first visit.

For the dietary assessment 24-hour dietary recalls will be applied in 3 different days. Subjects will be instructed not to change their dietary habits and to maintain their exercise levels during the length of the study.

Subject will visit the Research Center every two-weeks to receive a new bottle of pills and to answer an adherence questionnaire and also to ask for possible adverse events.

At week six in addition to the adherence questionnaire another blood sample and blood pressure will be taken. In addition, another 24-hour dietary recall will be completed

At the end of the 12 weeks all the basal assessments will be repeated.

Main study parameters/ endpoints Change from basal serum levels of the following parameters: measured basal and at the end of study: Carboxymethyl-lysine (CML), and sRAGE

Serum samples will be stored frozen at -80°C until assessment.

* Identification and quantification of CML will be measured with an immunoassay commercial kit (OxiSelect ™)
* Identification and quantification of sRAGE will be measured with Human RAGE Immunoassay commercial kit (Quantikine®)

Statistical analysis

Data will be presented as mean and standard deviation if presents normal distribution. Normality of data will be evaluated by Kolmogorov-Smirnov. To determinate basal differences between groups a t-Student test for independent samples will be applied. For the difference between groups before and after treatment a t-Student test for dependent samples will be applied. If data have not normal distribution, no parametrical tests will be used.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes:

* With no complications
* Not taking insulin
* With 5 years since diagnosis
* Not taking any vitamins
* Not pregnant or lactating women
* Not smoking

Exclusion Criteria:

* Intolerance to the benfotiamine treatment
* Lack of adherence (taking less than 80% of the pills)

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Serum levels of Carboxymethyl-lysine | 12 weeks
  Changes in serum levels of Carboxymethyl-lysine, a marker of AGEs, will be measured. Carboxymethyl-lysine serum levels will be measured by immunoassay and the units reported will be in milligrams per deciliter.

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Eugenia Garay-Sevilla, MD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Department of Medical Sciences, University of Guanajuato, León Mexico, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No